CLINICAL TRIAL: NCT02925533
Title: A Phase 1B Study of B-701 in Combination With Pembrolizumab in Relapsed or Refractory Locally Advanced or Metastatic Transitional Cell Carcinoma of the Urothelial Tract
Brief Title: Ph 1B B-701 in Combination With Pembrolizumab in Metastatic Transitional Cell Carcinoma of the Urothelial Tract
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to safety concerns.
Sponsor: Mark Pomerantz, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Rainier Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Mark Pomerantz, MD, Assistant Professor of Medicine, Harvard Medical School, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-246
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Urothelial Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — B701 protein, Human herpesvirus 6; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- B-701 and Pembrolizumab (Experimental): * B-701 will be administered every 3 weeks intravenously
  * Pembrolizumab will be administered every 3 weeks intravenously
  Interventions: Drug: B-701; Drug: Pembrolizumab

INTERVENTIONS:
Drug: B-701 — B-701 is a phage-derived, affinity-matured, human monoclonal antibody (mAb) specific for FGFR3. It is based on a human immunoglobulin G1 (IgG1) framework containing heavy chain VHIII and light chain VκI subgroup sequences.
Drug: Pembrolizumab — Pembrolizumab is an mAb that binds to the programmed cell death protein 1 (PD-1) receptor and blocks its interaction with programmed death-ligand 1 (PD-L1) and PD-L2, releasing PD-1 pathway-mediated inhibition of the immune response, including the anti-tumor immune response. In syngeneic mouse tumor models, blocking PD-1 activity resulted in decreased tumor growth.
  Other Names: Keytruda, MK-3475

SUMMARY:
This research study is studying a combination of two experimental drugs as a possible treatment for Bladder Cancer that recurred after treatment with standard therapy, or Bladder Cancer that got worse while on treatment with standard therapy.

The following interventions will be involved in this study:

* B-701
* Pembrolizumab

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved B-701 as a treatment for any disease.

The FDA has not approved Pembrolizumab for Bladder Cancer but it has been approved for other uses.

This is the first time that B-701 in combination with Pembrolizumab will be given to humans.

In this research study, Investigators are...

* Testing the effectiveness and safety of the combination of two experimental drugs (B-701 and Pembrolizumab);
* Learning about the good and/or bad effects the drugs have on participants and their cancer;
* Administering B-701 and Pembrolizumab, which are antibodies (proteins that bind to other molecules), because...

  * B-701 binds to a protein receptor called FGFR3 (fibroblast growth factor receptor 3). FGFR3 has been found to be present (expressed) or changed (mutated) on the surface of in many types of cancer cells. Targeting FGFR3 may inhibit cancer growth.
  * Pembrolizumab binds to a protein cell surface receptor called PD-1, which is found on certain types of lymphocytes and which are also involved in many types of cancer;
* Treating participants with Pembrolizumab, which is approved by the FDA for the treatment of Metastatic Melanoma, a Cancer of the skin;
* Collecting blood and tissue samples and other related medical information to learn more about the development of cancer and predictors of response;
* And hoping to learn how the combination of study drugs work in the treatment of cancer to help develop new treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have Stage IV, locally advanced or metastatic (T4b, any N; or any T, N2-3) urothelial bladder cancer or transitional cell carcinoma (TCC) arising in another location of the urinary tract, including urethra, ureter, and renal pelvis. The diagnosis must be histologically or cytologically confirmed. Mixed histologies are permitted as long as TCC is the major component (i.e. > 50% of the pathologic specimen). Pure or predominant squamous cell carcinomas or adenocarcinomas are not permitted.
* Relapsed after or refractory to one or two prior lines of chemotherapy for advanced or metastatic/recurrent disease (at least one cycle each) which have not included a PD-L1 or FGFR inhibitor. At least one regimen should have included a platinum agent unless contraindicated for the subject. Prior neoadjuvant or adjuvant chemotherapy (without a PD-L1 or FGFR inhibitor) is permitted and will not be counted as first-line chemotherapy, as long as the subject has not progressed within 12 months of the last dose. However, a regimen of neoadjuvant or adjuvant chemotherapy will be counted as first-line chemotherapy if the patient progressed within 12 months of the last dose.
* Age ≥ 18 years
* Eastern cooperative oncology group (ECOG) performance status ≤ 1 (Karnofsky ≥ 60%)
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥ 3000/mcL
  * absolute neutrophil count ≥ 1500/mcL
  * platelets ≥ 75,000/mcL
  * hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L
  * total bilirubin within normal institutional limits
  * EXCEPTION: Subjects with known Gilbert's disease: total bilirubin ≤ 3 × institutional upper limit of normal (ULN)
  * aspartate aminotransferase (AST) or serum glutamic oxaloacetic transaminase (SGOT)/Alanine aminotransferase (ALT) serum glutamic pyruvic transaminase (SGPT) ≤ 2.5 × institutional ULN
  * EXCEPTION: Subjects with documented liver metastases: AST and/or ALT ≤ 5 × institutional ULN
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥ 60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal (derived by the Cockcroft-Gault formula [Cockcroft 1976])
  * albumin ≥ 2.5 mg/dL
  * prothrombin time/international normalized ratio (PT/INR) and partial thromboplastin time (PTT) ≤ 1.5 × institutional ULN
* Note: Screening labs should be performed within 10 days of treatment initiation.
* Absence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule (such conditions should be discussed with the subject before study entry)
* The effects of B-701 on the developing human fetus are unknown. For this reason and because PD-1 inhibitors such as pembrolizumab may potentially cause fetal harm, women of child-bearing potential (defined as those who have not been surgically sterilized or have not been free from menses for > 1 year) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of study drug administration.
* Female of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medications. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study and through 4 months after the last dose of study medication.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who have had chemotherapy, targeted small molecule therapy, or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier.
* Participants who are receiving, or have received, any other investigational drugs or devices within the 2 weeks prior to the first dose of study medications.
* Participants who received major surgery must be recovered adequately from the toxicity and/or complications from the interventions prior to starting therapy.
* Participants with a diagnosis of immunodeficiency or who are receiving systemic steroid therapy (>5 mg prednisone or its equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
* Participants who have a primary central nervous system (CNS) malignancy, or untreated/active CNS metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control). Individuals with a history of treated CNS metastases are eligible, provided they meet all of the following criteria:

  * Evaluable or measurable disease outside the CNS
  * Radiographic demonstration of stability upon the completion of CNS directed therapy and no evidence of interim progression (for at least 4 weeks prior to the first dose of study drug) between the completion of CNS-directed therapy and the screening radiographic procedure
  * The screening CNS radiographic procedure is ≥ 8 weeks since completion of radiotherapy and ≥ 4 weeks since the discontinuation of corticosteroids and anticonvulsants Note: These exceptions do not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Participants with a history of allergic reactions attributed to monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
* Participants with active autoimmune disease that has required systemic treatment (>5 mg of prednisone or its equivalent) in the past 2 years (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Participants with known evidence of active, non-infectious pneumonitis.
* Participants with an active infection requiring systemic therapy.
* Participants who have received a live vaccine within 30 days of planned start of study therapy.

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

* Participants who have had a prior anti-cancer monoclonal antibody (mAb) within 2 weeks prior to Cycle 1 Day 1 or who have not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 2 weeks earlier.
* Participants unwilling or unable to discontinue use of prohibited therapies, including any cytotoxic chemotherapy, radiotherapy, immunotherapy or biologic agent (approved or investigational) for the treatment of TCC are ineligible.
* Participants with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participants who have undergone a major surgical procedure or trauma within 4 weeks prior to Cycle 1, Day 1. All wounds must be fully healed on Cycle 1, Day 1
* Participants with a history of other malignancy which could affect compliance with the protocol or interpretation of results. Individuals with a history of curatively treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix are allowed. Participants with a malignancy that has been treated with curative intent will also be allowed if the malignancy has been in remission without treatment for ≥ 2 years prior to Cycle 1, Day 1.
* Pregnant women are excluded from this study because the risks with B-701 are unknown and pembrolizumab is a PD-1 inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with B-701 and pembrolizumab, breastfeeding should be discontinued. Women of child-bearing potential must agree to use adequate birth control throughout the study duration.
* Hepatitis B, hepatitis C, and HIV serology-positive (or known history of HIV seropositive status) participants are ineligible because these underlying diseases will confound interpretation of important safety assessments, e.g. liver function tests, increased potential for reactivation or exacerbation of viral infections. Such individuals may be taking or require other drugs, and may be at higher risk of opportunistic infections and adverse effects. Hepatitis B, hepatitis C, and HIV serology-positive individuals were excluded from the pivotal pembrolizumab clinical trial in melanoma, so safety of this drug in this setting is unknown.
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at screening or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to Cycle 1, Day 1
* Has a known history of active TB (Bacillus Tuberculosis)
* Participants who weigh > 110 kg will be ineligible due to study drug limitations

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Preliminarily Evaluate The Safety Of B-701 In Combination With Pembrolizumab For The Treatment Of TCC | 2 years
  Safety will be assessed through summaries of AEs (adverse events), changes in laboratory test results, ECGs (electrocardiograms), and changes in vital signs

SECONDARY OUTCOMES:
To Assess The Efficacy Of B-701 In Combination With Pembrolizumab For The Treatment Of TCC | 2 years
  Measured by RECIST-based assessment of response and progression

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pomerantz, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No